CLINICAL TRIAL: NCT05853068
Title: Assessment of PaO2/FiO2 Ratio Pre and POst INTubation (The APPOINT Study)
Brief Title: Assessment of PaO2/FiO2 Ratio Pre and POst INTubation
Acronym: APPOINT
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jesus Villar, Principal investigator, Dr. Negrin University Hospital
Other Study IDs: 2022-161-1
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: acute respiratory failure; non-invasive ventilatory support; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients on non-invasive ventilatory support to IMV: Patients with AHRF treated with non-invasive ventilatory support [for the purpose of this study we included High-flow nasal cannula (HFNC), continuous positive airway pressure (CPAP), and non-invasive ventilation (NIV)] who required endotracheal intubation and invasive mechical ventilation.
  Interventions: Device: Mechanical ventilation

INTERVENTIONS:
Device: Mechanical ventilation — Need for endotracheal intubation and invasive mechanical ventilation

SUMMARY:
We designed this study to dtermine whether invasive mechanical ventilation (MV) would have an impact on the reclassification of patients with acute hypoxemic respiratory failure (AHRF) -treated previously with non-invasive respiratory support- into categories of severity (mild, moderate, and severe). Our hypothesis is that the assessment of PaO2/FiO2 ratio on PEEP greater or equal to 5 cmH2O after intubation, in patients labeled as mild/moderate/severe AHRF while on non-invasive respiratory support, would identify that a marked proportion of patients would change the degree of severity after a brief period of invasive MV

DETAILED DESCRIPTION:
Current criteria for definition of the acute respiratory distress syndrome (AHRF) are inadequate for inclusion of patients into clinical trials due to: (i) the lack of standardization for measuring the oxygenation defect (as assessed by the PaO2/FiO2 ratio) and (ii) the inclusion of non-intubated patients into the mild category of severity. We questioned whether the PaO2/FiO2 (P/F) ratio calculated before endotracheal intubation in non-intubated patients who otherwise meet AHRF criteria, would still meet the severity threshold once patients are intubated.

We will examine at 24 after intubation and initiation of MV whether adult patients with AHRF remained in the same AHRF category of severity (mild, moderate, severe) or do not meet the PaO2/FiO2 criterion for AHRF. If our hypothesis is supported, it would suggest that stratification of patients labeled based on P/F ratio while treated with non-invasive respiratory support is of limited utility for testing specific therapies for AHRF in non-intubated patients.

This is a high quality screening, longitudinal, defined population, retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting criteria for AHRF while they are on non-invasive respiratory support.
* We will only include patients who had arterial blood gases (ABG) within a time-frame of the last 5 hours of NIV and the first 5 hours of invasive MV.
* We will only include patients treated with high-flow oxygen nasal cannula (HFNC), or continuous positive airway pressure (CPAP), or bilevel positive pressure (BiPAP).

Exclusion Criteria:

* Patients who never required HFNC, or CPAP, or BiPAP before intubation.
* Patients with no ABG during the last 5 hours of NIV before intubation.
* Patients with no ABG during the first 5 hours after initiation of invasive MV.
* Patients treated with inhaled pulmonary vasodilator only before or only after intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AHRF (defined as PaO2/FiO2 lower or equal to 300 mmHg and FiO2 greater or equal to 0.3, on non-invasive ventilatory support) prior to intubation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the degree of lung severity | 60 days
  from severe/moderate to moderate/mild, from moderate/mild to mild after a brief period of invasive MV

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, Study Chair — Hospital Universitario D. Negrin
Locations (2):
- Rush University Medical Center, Chicago, Illinois, United States
- Jesús Villar, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No